CLINICAL TRIAL: NCT05615883
Title: Effects of Acute and Chronic Exercise on Myeloid-Derived Suppressor Cells in Melanoma Patients
Acronym: Agility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: INT 148/19; IG 2017 Project n. 20752 (Other Grant/Funding Number: AIRC)
Record Dates: First submitted 2021-04-29; First posted 2022-11-14 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2022-09

CONDITIONS: Melanoma
Keywords: Primary Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: Pre/post intervention, two-arms, sequential study. Patients with newly diagnose of melanoma are eligible.The study will enroll a total of 20 patients (10 in the AEP and 10 in the CEP), who will be enrolled approximately in 12-13 months.The first series of patients will be assigned to the Acute Exercise Program (AEP group), the second series to the Chronic Exercise Program (CEP group). The final endpoint is to verify whether short-term physical exercise can represent a feasible and safe tool for re-setting antitumor immunity in early melanoma patients. Investigators will analyze how the acute physical exercise modifies systemic immunity and biochemical/metabolic parameters. Specifically, Investigators will verify whether the exercise will modify:1 the immunological profiling of blood including frequency and function of MDSC, together with the concomitant status of antitumor immunity; 2 blood concentration of biochemical and metabolic parameters related to physical exercise and immunity
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AEP Group (Experimental): First series of patients (10 pts) will be assigned to the Acute Exercise Protocol Group (AEP Group). The acute program consists in a single walking session on a treadmill lasting 80 minutes. The exercise session will begin with a 10-minute warm-up at the patient's self selected comfortable speed. On the ending of warm up, treadmill speed will be increased until reaching target HRR zone. Then the treadmill speed will be maintained stable throughout the exercise session. Cardiac workload will be monitored by a Sport-watch (Garmin Forerunner) and the walking biomechanics by a foot sensor (Garmin Running Dynamic Pod Sensore).
  Interventions: Other: AEP Group Walking Sessions
- CEP Group (Experimental): Second series of patients (10 pts) will be assigned to the Chronic Exercise Protocol Group (CEP Group). The chronic program consists in a walking session on a treadmill lasting 80 minutes (depending on the AEP results), repeated three time a week for three weeks. The walking intensity will be defined during a treadmill test performedbefore the beginning of the exercise program. Each exercise session will beginwith a 10-minute warm-up at the patient's self selected comfortable speed. On the ending of warm up, patients will increase treadmill speed until reaching target HRR zone.Then the treadmill speed will be maintained stable throughout the exercise session. The first training session will be organized in hospital with supervision of research staff. Cardiac workload will be monitored by a Sport-watch (Garmin Forerunner) and walking biomechanics by a foot sensor (Garmin Running Dynamic Pod Sensore).
  Interventions: Other: CEP Group Walking Sessions

INTERVENTIONS:
Other: AEP Group Walking Sessions — The AEP Program consists in a single walking session on a treadmill lasting 80 minutes
  Arms: AEP Group
Other: CEP Group Walking Sessions — The chronic program consists in a walking session on a treadmill lasting 80 minutes (depending on the AEP results), repeated three time a week for three weeks.
  Arms: CEP Group

SUMMARY:
This study is designed to investigate the effects of ketogenic milieu induced by acute exercise as well as the effects of recurrent exercise bouts on functional status and the accumulation in peripheral blood of MDSCs and the consequent balance on antitumor immunity in melanoma patients.

DETAILED DESCRIPTION:
The screening period starts once a patient has provided written informed consent to participate in the study and ends on the day of exercise initiation. Screening assessments have to be done within 28 days prior to exercise initiation. The informed consent will adhere to IRB/ERC requirements, applicable laws and regulations. After the sign of an informed consensus, patients will be assigned to a specific exercise program. The first series of patients will be assigned to the Acute Exercise Program (AEP group), the second series to the Chronic Exercise Program (CEP group). The protocol will be implemented in the time between diagnosis and surgical intervention without any delay in the therapeutic pathway.

Basal evaluation: patient's life style will be investigated using the short version of Physical Activity Questionnaire (Italian version) and MeDiet questionnaire. Age, weight and eight will be registered for all patients. The Lean Body Mass will be measured by Dual Energy X-ray Absorptiometry (DEXA). A cardiorespiratory test will be performed to calculate an appropriate exercise intensity and subsequently the Six Minutes WalkingTest and the Comfortable Walking Speed test will be run before exercise protocol. In the CEP group the DEXA and the walking tests will be repeated after the end of exercise program.

Exercise prescription: the physical exercise consists in walking at a brisk pace. In order to produce a constant metabolic stress in patients with different aerobic power, walking intensity will be prescribed in accordance with the method of the Heart Rate Reserve (HRR), ie difference between resting heart rate (HR-resting) and the heart rate corresponding to muscle's maximal oxygen uptake (HR-max). This prescribing method is based on the linear relationship between heart rate reserve and muscle workload calculated as a percentage of the difference between resting and maximum muscle oxygen consumption (VO2R%). The training intensity will be set to the 30% HRR, the lowest intensity that produces a training effect. To minimize the impact of the research protocol on the patient's therapeutic path, the investigators refrain from the execution of a Cardio Pulmonary Exercise Test and therefore opted for calculating the HR-max using the ACSM formula. Given the entry criteria of this study the investigators believe this choice will minimally affect the exercise-dose prescription and study results.

Acute Exercise Protocol (AEP): The acute program consists in a single walking session on a treadmill lasting 80 minutes. The exercise session will begin with a 10-minute warm-up at the patient's self selected comfortable speed. On the ending of warm up, treadmill speed will be increased until reaching target HRR zone. Then the treadmill speed will be maintained stable throughout the exercise session. Cardiac workload will be monitored by a Sport-watch (Garmin Forerunner 35) and the walking biomechanics by a foot sensor (Garmin Running Dynamic Pod Sensore).

Chronic Exercise Protocol (CEP): The chronic program consists in a walking session on a treadmill lasting 80 minutes (depending on the AEP results), repeated three time a week for three weeks. The walking intensity will be defined during a treadmill test performed before the beginning of the exercise program. Each exercise session will begin with a 10-minute warm-up at the patient's self selected comfortable speed. On the ending of warm up, patients will increase treadmill speed until reaching target HRR zone. Then the treadmill speed will be maintained stable throughout the exercise session. The first training session will be organized in hospital with supervision of research staff. Cardiac workload will be monitored by a Sport-watch(Garmin Forerunner 35) and walking biomechanics by a foot sensor (Garmin Running Dynamic Pod Sensore).

Diet intervention: Modifications occurring during AEP strictly depend on the baseline metabolic conditions. For this reason, patients must remain fasting for 4 hours before the workout and avoid glucose rich foodies for 120 minutes after the end of exercise session in CEP group. During the exercise session patients will have free access to water only. All patients will complete a food diary during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years at the time of recruitment
* Histologically confirmed diagnosis of primary melanoma
* Patients who are candidate to curative surgery for primary melanoma, skin radicalization or sentinel node biopsy.
* American Society of Anaesthesiologists (ASA) status I
* Willingness and ability to comply with the protocol, the scheduled visits, treatment plans, laboratory tests and other procedures.
* Understanding and signature of the informed consent
* Female patients of childbearing potential must agree to sexual abstinence or to use highly effective method of contraception throughout the study (for CEP patients)

Exclusion Criteria:

* American Society of Anaesthesiologists (ASA) status > I
* Pregnancy or lactation
* Known infection from HIV virus
* Regular physical exercise (more than 1 exercise workout of moderate to intense exercise activity per week)
* Any physical or mental conditions interfering with the ability to perform exercise or to complete the testing procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Quantification of the immune cell subsets (to determine if occur the re-setting antitumor immunity by short-term physical exercise) | AEP group: before exercise session.
  Immune cells will be analyzed for frequency and function by 10-color flow cytometry to test the reciprocal balance of protumor vs antitumor immune subsets. The analysis, based in the application of multiple panels of different antibodies, will be performed on peripheral blood mononuclear cells (PBMC) isolated from peripheral blood.
Quantification of the immune cell subsets (to determine if occur the re-setting antitumor immunity by short-term physical exercise) | AEP group: after 40 minutes of exercise session.
  Immune cells will be analyzed for frequency and function by 10-color flow cytometry to test the reciprocal balance of protumor vs antitumor immune subsets. The analysis, based in the application of multiple panels of different antibodies, will be performed on peripheral blood mononuclear cells (PBMC) isolated from peripheral blood.
Quantification of the immune cell subsets (to determine if occur the re-setting antitumor immunity by short-term physical exercise) | AEP group: after 80 minutes of exercise session.
  Immune cells will be analyzed for frequency and function by 10-color flow cytometry to test the reciprocal balance of protumor vs antitumor immune subsets. The analysis, based in the application of multiple panels of different antibodies, will be performed on peripheral blood mononuclear cells (PBMC) isolated from peripheral blood.
Quantification of the immune cell subsets (to determine if occur the re-setting antitumor immunity by short-term physical exercise) | AEP group: at 24 post-exercise.
  Immune cells will be analyzed for frequency and function by 10-color flow cytometry to test the reciprocal balance of protumor vs antitumor immune subsets. The analysis, based in the application of multiple panels of different antibodies, will be performed on peripheral blood mononuclear cells (PBMC) isolated from peripheral blood.
Quantification of the immune cell subsets (to determine if occur the re-setting antitumor immunity by short-term physical exercise) | AEP group: at 72 hours post-exercise.
  Immune cells will be analyzed for frequency and function by 10-color flow cytometry to test the reciprocal balance of protumor vs antitumor immune subsets. The analysis, based in the application of multiple panels of different antibodies, will be performed on peripheral blood mononuclear cells (PBMC) isolated from peripheral blood.
Quantification of the immune cell subsets (to determine if occur the re-setting antitumor immunity by short-term physical exercise) | CEP group: before exercise program.
  Immune cells will be analyzed for frequency and function by 10-color flow cytometry to test the reciprocal balance of protumor vs antitumor immune subsets. The analysis, based in the application of multiple panels of different antibodies, will be performed on peripheral blood mononuclear cells (PBMC) isolated from peripheral blood.
Quantification of the immune cell subsets (to determine if occur the re-setting antitumor immunity by short-term physical exercise) | CEP group: after one week of exercise program.
  Immune cells will be analyzed for frequency and function by 10-color flow cytometry to test the reciprocal balance of protumor vs antitumor immune subsets. The analysis, based in the application of multiple panels of different antibodies, will be performed on peripheral blood mononuclear cells (PBMC) isolated from peripheral blood.
Quantification of the immune cell subsets (to determine if occur the re-setting antitumor immunity by short-term physical exercise) | CEP group: up to two weeks of exercise program.
  Immune cells will be analyzed for frequency and function by 10-color flow cytometry to test the reciprocal balance of protumor vs antitumor immune subsets. The analysis, based in the application of multiple panels of different antibodies, will be performed on peripheral blood mononuclear cells (PBMC) isolated from peripheral blood.
Transcriptional Immune cell profiling (to determine if occur the re-setting antitumor immunity by short-term physical exercise) | AEP group: before exercise.
  CD14+, CD15+ and total immune cells will be immunosorted directly from whole blood (3 ml) and frozen for the targeted expression profiling of signaling pathways and functional patterns (Nanostring or customized PCR cards).
Transcriptional Immune cell profiling (to determine if occur the re-setting antitumor immunity by short-term physical exercise) | AEP group: after 40 minutes of exercise session
  CD14+, CD15+ and total immune cells will be immunosorted directly from whole blood (3 ml) and frozen for the targeted expression profiling of signaling pathways and functional patterns (Nanostring or customized PCR cards).
Transcriptional Immune cell profiling (to determine if occur the re-setting antitumor immunity by short-term physical exercise) | AEP group: after 80 minutes of exercise session.
  CD14+, CD15+ and total immune cells will be immunosorted directly from whole blood (3 ml) and frozen for the targeted expression profiling of signaling pathways and functional patterns (Nanostring or customized PCR cards).
Transcriptional Immune cell profiling (to determine if occur the re-setting antitumor immunity by short-term physical exercise) | AEP group: at 24 post-exercise.
  CD14+, CD15+ and total immune cells will be immunosorted directly from whole blood (3 ml) and frozen for the targeted expression profiling of signaling pathways and functional patterns (Nanostring or customized PCR cards).
Transcriptional Immune cell profiling (to determine if occur the re-setting antitumor immunity by short-term physical exercise) | AEP group: at 72 hours post-exercise.
  CD14+, CD15+ and total immune cells will be immunosorted directly from whole blood (3 ml) and frozen for the targeted expression profiling of signaling pathways and functional patterns (Nanostring or customized PCR cards).
Transcriptional Immune cell profiling (to determine if occur the re-setting antitumor immunity by short-term physical exercise) | CEP group: before exercise program.
  CD14+, CD15+ and total immune cells will be immunosorted directly from whole blood (3 ml) and frozen for the targeted expression profiling of signaling pathways and functional patterns (Nanostring or customized PCR cards).
Transcriptional Immune cell profiling (to determine if occur the re-setting antitumor immunity by short-term physical exercise) | CEP group: after one week of exercise program.
  CD14+, CD15+ and total immune cells will be immunosorted directly from whole blood (3 ml) and frozen for the targeted expression profiling of signaling pathways and functional patterns (Nanostring or customized PCR cards).
Transcriptional Immune cell profiling (to determine if occur the re-setting antitumor immunity by short-term physical exercise) | CEP group: up to two weeks of exercise program.
  CD14+, CD15+ and total immune cells will be immunosorted directly from whole blood (3 ml) and frozen for the targeted expression profiling of signaling pathways and functional patterns (Nanostring or customized PCR cards).
Analysis of the "systemic metabolic milieu"_AEPMet before | AEP group: before exercise.
  In plasma we will quantify pH, Lactate, Ketone bodies, Free Fatty Acids, Glucose and Insulin serum levels that will be combined to report the metabolic parameters
Analysis of the "systemic metabolic milieu"_AEPHor before | AEP group: before exercise.
  In serum we will quantify ACTH, cortisol, epinephrine and norepinephrine concentrations that will be combined to report the hormonal parameters
Analysis of the "systemic metabolic milieu"_AEPInf before | AEP group: before exercise.
  In blood we will quantify IL-6, CRP, inflammatory cito/chemokines such as IL8, CCL2, IFN, IL10, IL1b, TNFa, TGFb that will be combined to report the inflammatory parameters
Analysis of the "systemic metabolic milieu"_AEPLip before | AEP group: before exercise.
  We will analyze the Lipidomics and amino acid profiles by laboratory test that will be combined to report the composition of cell membranes
Analysis of the "systemic metabolic milieu"_AEPcounts before | AEP group: before exercise.
  Whole blood cell counts will be also performed; this parameter is characterized by the absolute number as well as relative ratio.
Analysis of the "systemic metabolic milieu"_AEPMet 40 | AEP group: after 40 minutes of exercise session.
  In plasma we will quantify pH, Lactate, Ketone bodies, Free Fatty Acids, Glucose and Insulin serum levels that will be combined to report the metabolic parameters
Analysis of the "systemic metabolic milieu"_AEPHor 40 | AEP group: after 40 minutes of exercise session.
  In serum we will quantify ACTH, cortisol, epinephrine and norepinephrine concentrations that will be combined to report the hormonal parameters
Analysis of the "systemic metabolic milieu"_AEPInf 40 | AEP group: after 40 minutes of exercise session.
  In blood we will quantify IL-6, CRP, inflammatory cito/chemokines such as IL8, CCL2, IFN, IL10, IL1b, TNFa, TGFb that will be combined to report the inflammatory parameters
Analysis of the "systemic metabolic milieu"_AEPLip 40 | AEP group: after 40 minutes of exercise session.
  We will analyze the Lipidomics and amino acid profiles by laboratory test that will be combined to report the composition of cell membranes
Analysis of the "systemic metabolic milieu"_AEPcounts 40 | AEP group: after 40 minutes of exercise session.
  Whole blood cell counts will be also performed; this parameter is characterized by the absolute number as well as relative ratio.
Analysis of the "systemic metabolic milieu"_AEPMet 80 | AEP group: after 80 minutes of exercise session.
  In plasma we will quantify pH, Lactate, Ketone bodies, Free Fatty Acids, Glucose and Insulin serum levels that will be combined to report the metabolic parameters
Analysis of the "systemic metabolic milieu"_AEPHor 80 | AEP group: after 80 minutes of exercise session.
  In serum we will quantify ACTH, cortisol, epinephrine and norepinephrine concentrations that will be combined to report the hormonal parameters
Analysis of the "systemic metabolic milieu"_AEPInf 80 | AEP group: after 80 minutes of exercise session.
  In blood we will quantify IL-6, CRP, inflammatory cito/chemokines such as IL8, CCL2, IFN, IL10, IL1b, TNFa, TGFb that will be combined to report the inflammatory parameters
Analysis of the "systemic metabolic milieu"_AEPLip 80 | AEP group: after 80 minutes of exercise session.
  We will analyze the Lipidomics and amino acid profiles by laboratory test that will be combined to report the composition of cell membranes
Analysis of the "systemic metabolic milieu"_AEPcounts 80 | AEP group: after 80 minutes of exercise session.
  Whole blood cell counts will be also performed; this parameter is characterized by the absolute number as well as relative ratio.
Analysis of the "systemic metabolic milieu"_AEPMet 24 | AEP group: at 24 post-exercise.
  In plasma we will quantify pH, Lactate, Ketone bodies, Free Fatty Acids, Glucose and Insulin serum levels that will be combined to report the metabolic parameters
Analysis of the "systemic metabolic milieu"_AEPHor 24 | AEP group: at 24 post-exercise.
  In serum we will quantify ACTH, cortisol, epinephrine and norepinephrine concentrations that will be combined to report the hormonal parameters
Analysis of the "systemic metabolic milieu"_AEPInf 24 | AEP group: at 24 post-exercise.
  In blood we will quantify IL-6, CRP, inflammatory cito/chemokines such as IL8, CCL2, IFN, IL10, IL1b, TNFa, TGFb that will be combined to report the inflammatory parameters
Analysis of the "systemic metabolic milieu"_AEPLip 24 | AEP group: at 24 post-exercise.
  We will analyze the Lipidomics and amino acid profiles by laboratory test that will be combined to report the composition of cell membranes
Analysis of the "systemic metabolic milieu"_AEPcounts 24 | AEP group: at 24 post-exercise.
  Whole blood cell counts will be also performed; this parameter is characterized by the absolute number as well as relative ratio.
Analysis of the "systemic metabolic milieu"_AEPMet 72 | AEP group: at 72 hours post-exercise.
  In plasma we will quantify pH, Lactate, Ketone bodies, Free Fatty Acids, Glucose and Insulin serum levels that will be combined to report the metabolic parameters
Analysis of the "systemic metabolic milieu"_AEPHor 72 | AEP group: at 72 hours post-exercise.
  In serum we will quantify ACTH, cortisol, epinephrine and norepinephrine concentrations that will be combined to report the hormonal parameters
Analysis of the "systemic metabolic milieu"_AEPInf 72 | AEP group: at 72 hours post-exercise.
  In blood we will quantify IL-6, CRP, inflammatory cito/chemokines such as IL8, CCL2, IFN, IL10, IL1b, TNFa, TGFb that will be combined to report the inflammatory parameters
Analysis of the "systemic metabolic milieu"_AEPLip 72 | AEP group: at 72 hours post-exercise.
  We will analyze the Lipidomics and amino acid profiles by laboratory test that will be combined to report the composition of cell membranes
Analysis of the "systemic metabolic milieu"_AEPcounts 72 | AEP group: at 72 hours post-exercise.
  Whole blood cell counts will be also performed; this parameter is characterized by the absolute number as well as relative ratio.
Analysis of the "systemic metabolic milieu"_CEPMet before | CEP group: before exercise program.
  In plasma we will quantify pH, Lactate, Ketone bodies, Free Fatty Acids, Glucose and Insulin serum levels that will be combined to report the metabolic parameters
Analysis of the "systemic metabolic milieu"_CEPHor before | CEP group: before exercise program.
  In serum we will quantify ACTH, cortisol, epinephrine and norepinephrine concentrations that will be combined to report the hormonal parameters
Analysis of the "systemic metabolic milieu"_CEPInf before | CEP group: before exercise program.
  In blood we will quantify IL-6, CRP, inflammatory cito/chemokines such as IL8, CCL2, IFN, IL10, IL1b, TNFa, TGFb that will be combined to report the inflammatory parameters
Analysis of the "systemic metabolic milieu"_CEPLip before | CEP group: before exercise program.
  We will analyze the Lipidomics and amino acid profiles by laboratory test that will be combined to report the composition of cell membranes
Analysis of the "systemic metabolic milieu"_CEP counts before | CEP group: before exercise program.
  Whole blood cell counts will be also performed; this parameter is characterized by the absolute number as well as relative ratio.
Analysis of the "systemic metabolic milieu"_CEPMet 1w | CEP group: after one week of exercise program.
  In plasma we will quantify pH, Lactate, Ketone bodies, Free Fatty Acids, Glucose and Insulin serum levels that will be combined to report the metabolic parameters
Analysis of the "systemic metabolic milieu"_CEPHor 1w | CEP group: after one week of exercise program.
  In serum we will quantify ACTH, cortisol, epinephrine and norepinephrine concentrations that will be combined to report the hormonal parameters
Analysis of the "systemic metabolic milieu"_CEPInf 1w | CEP group: after one week of exercise program.
  In blood we will quantify IL-6, CRP, inflammatory cito/chemokines such as IL8, CCL2, IFN, IL10, IL1b, TNFa, TGFb that will be combined to report the inflammatory parameters
Analysis of the "systemic metabolic milieu"_CEPLip 1w | CEP group: after one week of exercise program.
  We will analyze the Lipidomics and amino acid profiles by laboratory test that will be combined to report the composition of cell membranes
Analysis of the "systemic metabolic milieu"_CEPcounts 1w | CEP group: after one week of exercise program.
  Whole blood cell counts will be also performed; this parameter is characterized by the absolute number as well as relative ratio.
Analysis of the "systemic metabolic milieu"_CEPMet 2w | CEP group: up to two week of exercise program.
  In plasma we will quantify pH, Lactate, Ketone bodies, Free Fatty Acids, Glucose and Insulin serum levels that will be combined to report the metabolic parameters
Analysis of the "systemic metabolic milieu"_CEPHor 2w | CEP group: up to two week of exercise program.
  In serum we will quantify ACTH, cortisol, epinephrine and norepinephrine concentrations that will be combined to report the hormonal parameters
Analysis of the "systemic metabolic milieu"_CEPInf 2w | CEP group: up to two week of exercise program.
  In blood we will quantify IL-6, CRP, inflammatory cito/chemokines such as IL8, CCL2, IFN, IL10, IL1b, TNFa, TGFb that will be combined to report the inflammatory parameters
Analysis of the "systemic metabolic milieu"_CEPLip 2w | CEP group: up to two week of exercise program.
  We will analyze the Lipidomics and amino acid profiles by laboratory test that will be combined to report the composition of cell membranes
Analysis of the "systemic metabolic milieu"_CEPcounts 2w | CEP group: up to two week of exercise program.
  Whole blood cell counts will be also performed; this parameter is characterized by the absolute number as well as relative ratio.
Analysis of the metabolic parameters by capillary sampling_AEPCap before | AEP group: before exercise session.
  Capillary sampling (prick sampling) to analysis metabolic parameters at systemic blood level will be performed during the first, in-hospital, training session and further will be continued at home, self-managed by the patient who will have to measure glycaemia and ketones every morning (finger prick sampling) and after each training sessions (earlobe prick sampling).
Analysis of the metabolic parameters by capillary sampling_AEPCap 40 | AEP group: after 40 minutes of exercise session.
  Capillary sampling (prick sampling) to analysis metabolic parameters at systemic blood level will be performed during the first, in-hospital, training session and further will be continued at home, self-managed by the patient who will have to measure glycaemia and ketones every morning (finger prick sampling) and after each training sessions (earlobe prick sampling).
Analysis of the metabolic parameters by capillary sampling_AEPCap 80 | AEP group: after 80 minutes of exercise session.
  Capillary sampling (prick sampling) to analysis metabolic parameters at systemic blood level will be performed during the first, in-hospital, training session and further will be continued at home, self-managed by the patient who will have to measure glycaemia and ketones every morning (finger prick sampling) and after each training sessions (earlobe prick sampling).
Analysis of the metabolic parameters by capillary sampling_AEPCap 24 | AEP group: at 24 post-exercise.
  Capillary sampling (prick sampling) to analysis metabolic parameters at systemic blood level will be performed during the first, in-hospital, training session and further will be continued at home, self-managed by the patient who will have to measure glycaemia and ketones every morning (finger prick sampling) and after each training sessions (earlobe prick sampling).
Analysis of the metabolic parameters by capillary sampling_AEPCap 72 | AEP group: at 72 hours post-exercise.
  Capillary sampling (prick sampling) to analysis metabolic parameters at systemic blood level will be performed during the first, in-hospital, training session and further will be continued at home, self-managed by the patient who will have to measure glycaemia and ketones every morning (finger prick sampling) and after each training sessions (earlobe prick sampling).
Analysis of the metabolic parameters by capillary sampling_CEPCap before | CEP group: during the first training session
  Capillary sampling (prick sampling) to analysis metabolic parameters at systemic blood level will be performed during the first, in-hospital, training session and further will be continued at home, self-managed by the patient who will have to measure glycaemia and ketones every morning (finger prick sampling) and after each training sessions (earlobe prick sampling).
Analysis of the metabolic parameters by capillary sampling_CEPCap 2w | CEP group: every morning up to two weeks.
  Capillary sampling (prick sampling) to analysis metabolic parameters at systemic blood level will be performed during the first, in-hospital, training session and further will be continued at home, self-managed by the patient who will have to measure glycaemia and ketones every morning (finger prick sampling) and after each training sessions (earlobe prick sampling).
Analysis of the metabolic parameters by capillary sampling_CEPCap end | CEP group: at the end of training sessions up to two weeks.
  Capillary sampling (prick sampling) to analysis metabolic parameters at systemic blood level will be performed during the first, in-hospital, training session and further will be continued at home, self-managed by the patient who will have to measure glycaemia and ketones every morning (finger prick sampling) and after each training sessions (earlobe prick sampling).

OTHER OUTCOMES:
Physical Activity Questionnaire | Within one month of the enrollment
  Patient's life style will be investigated using the short version of Physical Activity Questionnaire
MeDiet questionnaire | Within one month of the enrollment
  Patient's life style will be investigated using the short version of MeDiet questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Licia Rivoltini, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano, Italy
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
Since the study data could be compared with those obtained from other clinical studies, focused on the immune system, this part is not yet defined. Anyhow it will depend on the results obtained.

REFERENCES:
- [Background] Yuan HX, Xiong Y, Guan KL. Nutrient sensing, metabolism, and cell growth control. Mol Cell. 2013 Feb 7;49(3):379-87. doi: 10.1016/j.molcel.2013.01.019. PMID 23395268
- [Background] Dazert E, Hall MN. mTOR signaling in disease. Curr Opin Cell Biol. 2011 Dec;23(6):744-55. doi: 10.1016/j.ceb.2011.09.003. Epub 2011 Sep 29. PMID 21963299
- [Background] Buck MD, Sowell RT, Kaech SM, Pearce EL. Metabolic Instruction of Immunity. Cell. 2017 May 4;169(4):570-586. doi: 10.1016/j.cell.2017.04.004. PMID 28475890
- [Background] Biswas SK. Metabolic Reprogramming of Immune Cells in Cancer Progression. Immunity. 2015 Sep 15;43(3):435-49. doi: 10.1016/j.immuni.2015.09.001. PMID 26377897
- [Background] Longo VD, Mattson MP. Fasting: molecular mechanisms and clinical applications. Cell Metab. 2014 Feb 4;19(2):181-92. doi: 10.1016/j.cmet.2013.12.008. Epub 2014 Jan 16. PMID 24440038
- [Background] Filipazzi P, Huber V, Rivoltini L. Phenotype, function and clinical implications of myeloid-derived suppressor cells in cancer patients. Cancer Immunol Immunother. 2012 Feb;61(2):255-263. doi: 10.1007/s00262-011-1161-9. Epub 2011 Nov 27. PMID 22120756
- [Background] Jian SL, Chen WW, Su YC, Su YW, Chuang TH, Hsu SC, Huang LR. Glycolysis regulates the expansion of myeloid-derived suppressor cells in tumor-bearing hosts through prevention of ROS-mediated apoptosis. Cell Death Dis. 2017 May 11;8(5):e2779. doi: 10.1038/cddis.2017.192. PMID 28492541
- [Background] Trikha P, Plews RL, Stiff A, Gautam S, Hsu V, Abood D, Wesolowski R, Landi I, Mo X, Phay J, Chen CS, Byrd J, Caligiuri M, Tridandapani S, Carson W. Targeting myeloid-derived suppressor cells using a novel adenosine monophosphate-activated protein kinase (AMPK) activator. Oncoimmunology. 2016 Jul 25;5(9):e1214787. doi: 10.1080/2162402X.2016.1214787. eCollection 2016. PMID 27757311
- [Background] Li W, Tanikawa T, Kryczek I, Xia H, Li G, Wu K, Wei S, Zhao L, Vatan L, Wen B, Shu P, Sun D, Kleer C, Wicha M, Sabel M, Tao K, Wang G, Zou W. Aerobic Glycolysis Controls Myeloid-Derived Suppressor Cells and Tumor Immunity via a Specific CEBPB Isoform in Triple-Negative Breast Cancer. Cell Metab. 2018 Jul 3;28(1):87-103.e6. doi: 10.1016/j.cmet.2018.04.022. Epub 2018 May 24. PMID 29805099
- [Background] Ball D. Metabolic and endocrine response to exercise: sympathoadrenal integration with skeletal muscle. J Endocrinol. 2015 Feb;224(2):R79-95. doi: 10.1530/JOE-14-0408. Epub 2014 Nov 27. PMID 25431226
- [Background] Pedersen BK, Febbraio MA. Muscle as an endocrine organ: focus on muscle-derived interleukin-6. Physiol Rev. 2008 Oct;88(4):1379-406. doi: 10.1152/physrev.90100.2007. PMID 18923185
- [Background] Wasserman DH. Four grams of glucose. Am J Physiol Endocrinol Metab. 2009 Jan;296(1):E11-21. doi: 10.1152/ajpendo.90563.2008. Epub 2008 Oct 7. PMID 18840763
- [Background] Murray B, Rosenbloom C. Fundamentals of glycogen metabolism for coaches and athletes. Nutr Rev. 2018 Apr 1;76(4):243-259. doi: 10.1093/nutrit/nuy001. PMID 29444266
- [Background] Purdom T, Kravitz L, Dokladny K, Mermier C. Understanding the factors that effect maximal fat oxidation. J Int Soc Sports Nutr. 2018 Jan 12;15:3. doi: 10.1186/s12970-018-0207-1. eCollection 2018. PMID 29344008
- [Background] Brooks GA, Mercier J. Balance of carbohydrate and lipid utilization during exercise: the "crossover" concept. J Appl Physiol (1985). 1994 Jun;76(6):2253-61. doi: 10.1152/jappl.1994.76.6.2253. PMID 7928844
- [Background] Goodwin ML. Blood glucose regulation during prolonged, submaximal, continuous exercise: a guide for clinicians. J Diabetes Sci Technol. 2010 May 1;4(3):694-705. doi: 10.1177/193229681000400325. PMID 20513337
- [Background] Puchalska P, Crawford PA. Multi-dimensional Roles of Ketone Bodies in Fuel Metabolism, Signaling, and Therapeutics. Cell Metab. 2017 Feb 7;25(2):262-284. doi: 10.1016/j.cmet.2016.12.022. PMID 28178565
- [Background] Evans M, Cogan KE, Egan B. Metabolism of ketone bodies during exercise and training: physiological basis for exogenous supplementation. J Physiol. 2017 May 1;595(9):2857-2871. doi: 10.1113/JP273185. Epub 2016 Dec 7. PMID 27861911
- [Background] Fisher JS, Gao J, Han DH, Holloszy JO, Nolte LA. Activation of AMP kinase enhances sensitivity of muscle glucose transport to insulin. Am J Physiol Endocrinol Metab. 2002 Jan;282(1):E18-23. doi: 10.1152/ajpendo.2002.282.1.E18. PMID 11739078
- [Background] Geiger PC, Wright DC, Han DH, Holloszy JO. Activation of p38 MAP kinase enhances sensitivity of muscle glucose transport to insulin. Am J Physiol Endocrinol Metab. 2005 Apr;288(4):E782-8. doi: 10.1152/ajpendo.00477.2004. Epub 2004 Dec 7. PMID 15585585
- [Background] Sawanobori Y, Ueha S, Kurachi M, Shimaoka T, Talmadge JE, Abe J, Shono Y, Kitabatake M, Kakimi K, Mukaida N, Matsushima K. Chemokine-mediated rapid turnover of myeloid-derived suppressor cells in tumor-bearing mice. Blood. 2008 Jun 15;111(12):5457-66. doi: 10.1182/blood-2008-01-136895. Epub 2008 Mar 28. PMID 18375791
- [Background] Condamine T, Kumar V, Ramachandran IR, Youn JI, Celis E, Finnberg N, El-Deiry WS, Winograd R, Vonderheide RH, English NR, Knight SC, Yagita H, McCaffrey JC, Antonia S, Hockstein N, Witt R, Masters G, Bauer T, Gabrilovich DI. ER stress regulates myeloid-derived suppressor cell fate through TRAIL-R-mediated apoptosis. J Clin Invest. 2014 Jun;124(6):2626-39. doi: 10.1172/JCI74056. Epub 2014 May 1. PMID 24789911
- [Background] Motallebnezhad M, Jadidi-Niaragh F, Qamsari ES, Bagheri S, Gharibi T, Yousefi M. The immunobiology of myeloid-derived suppressor cells in cancer. Tumour Biol. 2016 Feb;37(2):1387-406. doi: 10.1007/s13277-015-4477-9. Epub 2015 Nov 26. PMID 26611648
- [Background] Khaled YS, Ammori BJ, Elkord E. Myeloid-derived suppressor cells in cancer: recent progress and prospects. Immunol Cell Biol. 2013 Sep;91(8):493-502. doi: 10.1038/icb.2013.29. Epub 2013 Jun 25. PMID 23797066
- [Background] Psaila B, Lyden D. The metastatic niche: adapting the foreign soil. Nat Rev Cancer. 2009 Apr;9(4):285-93. doi: 10.1038/nrc2621. PMID 19308068
- [Background] Umansky V, Sevko A, Gebhardt C, Utikal J. Myeloid-derived suppressor cells in malignant melanoma. J Dtsch Dermatol Ges. 2014 Nov;12(11):1021-7. doi: 10.1111/ddg.12411. Epub 2014 Sep 28. English, German. PMID 25263083
- [Background] Carruba G, Cocciadiferro L, Di Cristina A, Granata OM, Dolcemascolo C, Campisi I, Zarcone M, Cinquegrani M, Traina A. Nutrition, aging and cancer: lessons from dietary intervention studies. Immun Ageing. 2016 Apr 7;13:13. doi: 10.1186/s12979-016-0069-9. eCollection 2016. PMID 27057203
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] McCulloch KL, Mercer V, Giuliani C, Marshall S. Development of a clinical measure of dual-task performance in walking: reliability and preliminary validity of the Walking and Remembering Test. J Geriatr Phys Ther. 2009;32(1):2-9. doi: 10.1519/00139143-200932010-00002. PMID 19856629
- [Background] da Cunha FA, Farinatti Pde T, Midgley AW. Methodological and practical application issues in exercise prescription using the heart rate reserve and oxygen uptake reserve methods. J Sci Med Sport. 2011 Jan;14(1):46-57. doi: 10.1016/j.jsams.2010.07.008. Epub 2010 Sep 15. PMID 20833587
- [Background] Mann T, Lamberts RP, Lambert MI. Methods of prescribing relative exercise intensity: physiological and practical considerations. Sports Med. 2013 Jul;43(7):613-25. doi: 10.1007/s40279-013-0045-x. PMID 23620244
- [Background] Swain DP, Franklin BA. VO(2) reserve and the minimal intensity for improving cardiorespiratory fitness. Med Sci Sports Exerc. 2002 Jan;34(1):152-7. doi: 10.1097/00005768-200201000-00023. PMID 11782661
- [Background] Tanaka H, Monahan KD, Seals DR. Age-predicted maximal heart rate revisited. J Am Coll Cardiol. 2001 Jan;37(1):153-6. doi: 10.1016/s0735-1097(00)01054-8. PMID 11153730